CLINICAL TRIAL: NCT04145089
Title: Comparative Study of Time Taken for Intubation and Cormack Lehane View Between C-Mac Video Laryngoscopy With Glidescope Video Laryngoscopy in Paediatric Patients Undergoing Elective Surgery
Brief Title: Comparison of Time Taken for Intubation and Cormack Lehane View Between C-Mac With Glidescope Video Laryngoscopy in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: FF-2019-004
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-09

CONDITIONS: Paediatric Airway

STUDY DESIGN:
Intervention Model Description: GlideScope intubation Vs Cmac intubation
Who Masked: Participant
Masking Description: Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-Mac intubation (Active Comparator): Intubation with C-MAC video laryngoscopy
  Interventions: Device: Glidescope video laryngoscopy/ C-MAC video laryngoscopy
- Glidescope intubation (Active Comparator): Intubation with Glidescope video laryngoscopy
  Interventions: Device: Glidescope video laryngoscopy/ C-MAC video laryngoscopy

INTERVENTIONS:
Device: Glidescope video laryngoscopy/ C-MAC video laryngoscopy — usage of said devices according to manual

SUMMARY:
This study compares the time taken to intubate between Cmac video laryngoscopy with Glidescope video laryngoscopy in paediatric patients aged 3-12 years old.

DETAILED DESCRIPTION:
This study aims to determine whether are both devices comparable to each other in terms of intubation time and Cormack Lehane view in paediatric patients with normal airway undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients 3-12 years old undergoing elective surgery
* American Society of Anesthesiology (ASA) 1-2
* No difficult airway features/history of difficult intubation
* Not obese

Exclusion Criteria:

* Any difficult intubation features/history of difficult intubation
* Obese child

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Intubation time | 5 minutes
  Time taken from insertion of specified laryngoscope blade to lip until presence of capnography tracing

SECONDARY OUTCOMES:
Cormack Lehane view | 5 minutes
  grade from 1-4 by operator's assesment

OTHER OUTCOMES:
Additional maneuvre to assist intubation | 5 minutes
  i.e external laryngeal manipulation, bougie assisted
adverse events | 5 minutes
  i.e lip injury, desaturations

CONTACTS AND LOCATIONS:
Overall Officials: Syarifah Noor Nazihah Sayed Masri, MD, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holm-Knudsen RJ, Rasmussen LS. Paediatric airway management: basic aspects. Acta Anaesthesiol Scand. 2009 Jan;53(1):1-9. doi: 10.1111/j.1399-6576.2008.01794.x. PMID 19128325
- [Background] Armstrong J, John J, Karsli C. A comparison between the GlideScope Video Laryngoscope and direct laryngoscope in paediatric patients with difficult airways - a pilot study. Anaesthesia. 2010 Apr;65(4):353-7. doi: 10.1111/j.1365-2044.2010.06294.x. PMID 20402873
- [Background] Mosier J, Chiu S, Patanwala AE, Sakles JC. A comparison of the GlideScope video laryngoscope to the C-MAC video laryngoscope for intubation in the emergency department. Ann Emerg Med. 2013 Apr;61(4):414-420.e1. doi: 10.1016/j.annemergmed.2012.11.001. Epub 2013 Jan 30. PMID 23374414
- [Background] Hurford DM, White MC. A comparison of the Glidescope and Karl Storz DCI videolaryngoscopes in a paediatric manikin. Anaesthesia. 2010 Aug;65(8):781-4. doi: 10.1111/j.1365-2044.2010.06390.x. Epub 2010 Jun 2. PMID 20528838
- [Background] Kim JT, Na HS, Bae JY, Kim DW, Kim HS, Kim CS, Kim SD. GlideScope video laryngoscope: a randomized clinical trial in 203 paediatric patients. Br J Anaesth. 2008 Oct;101(4):531-4. doi: 10.1093/bja/aen234. Epub 2008 Aug 8. PMID 18689807